CLINICAL TRIAL: NCT03822650
Title: A Natural History and Outcome Measure Discovery Study of Neuronal Ceroid Lipofuscinosis Type 5 (CLN5)
Brief Title: A Natural History Study of Neuronal Ceroid Lipofuscinosis Type 5 (CLN5)
Status: Completed | Type: Observational
Sponsor: Neurogene Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-100
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Ceroid Lipofuscinosis, Neuronal 5
Keywords: CLN; NCL; Batten
MeSH Terms: conditions — Ceroid lipofuscinosis, neuronal 5

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective: Subjects who meet eligibility criteria and enroll in the prospective arm will be assessed every 6 months ± 4 weeks for a period of up to 3 years, according to the Schedule of Assessments.
  Subjects in the Prospective arm may also participate in the Retrospective arm.
- Retrospective: Upon confirmation of eligibility criteria, the site will obtain an Informed Consent/Assent form and release of medical records from the subject/legally authorized representative to allow review of the medical records from the subject's primary care physician and/or specialists to confirm the CLN5 diagnosis and disease course. To facilitate collection of the medical records, a caregiver interview will be completed at initial enrollment then once yearly for up to 3 years.

SUMMARY:
CLN5 is a form of Batten Disease, a neurodegenerative disorder in children causing psychomotor regression, seizures, blindness, loss of ambulation and premature death, and has no available treatments.

The purpose of this study is to investigate the clinical characteristics and natural clinical progression of symptoms in individuals with CLN5. This natural history study is important to better understand disease course to be able to determine clinically relevant outcome measures for use in future clinical trials.

DETAILED DESCRIPTION:
Neuronal Ceroid Lipofuscinosis (NCL) are comprised of a group of fatal neurodegenerative diseases caused by mutations in an enzyme or protein which results in the accumulation of toxic deposits in the eye, brain, skin, muscle and other cells.

CLN5 is a type of NCL, caused by homozygous or bi-allelic heterozygous variants in the CLN5 gene. Lack of CLN5 protein impairs the breakdown of certain proteins, leads to defective lysosomal trafficking, resulting in accumulation of toxic material and subsequent cell damage. CLN5 disease presents in childhood with neurological findings including motor clumsiness and attention disturbances, followed by progressive visual failure, psychomotor depression, epilepsy, and premature death.

No investigational product will be provided in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age at disease onset of ≤ 5 years of age.
2. Molecular genetic diagnosis confirming the presence of pathogenic or likely pathogenic variant(s) on both alleles (biallelic) of the CLN5 gene.

For Prospective Arm only:

1. Subject age of ≤ 9 years.
2. Hamburg motor and vision score of ≥ 1 at time of consent.
3. Subject must have a caregiver available to support the subject and attend visits with the subject.

Exclusion Criteria - All Subjects:

1. Has another neurologic disease or illness that may have caused cognitive decline before study entry.
2. Has a known pathogenic or clinically suspected mutation in a seizure associated genetic mutation besides CLN5.
3. Any prior participation in a study in which a gene therapy vector or stem cell transplantation was administered.
4. Participation in other investigational studies and non-interventional studies that have similar study assessments as this protocol while the subject is enrolled in this study is prohibited.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed genetic diagnosis of CLN5.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Unified Batten Disease Rating Scale (UBDRS) | 3 years
  Disease-specific clinical assessment used to assess physical, seizure, behavioral and functional capabilities. For physical assessments scores range from 0 to 4 with the score of 4 being most severe.
Late Infantile Neuronal Ceroid Lipofuscinosis Rating Scale (Hamburg Scale) | 3 years
  Disease specific tool used to capture 4 domains including motor function, seizures, visual function and language. Each sub-scale can be scored from 0-3 points in which 0 represents loss of function.

SECONDARY OUTCOMES:
Electroencephalography (EEG) | 3 years
  EEG records electrical brain activity and Interictal discharges (location, focal/generalized, etc) will be compared to baseline and characterized over time.
Vineland Adaptive Behavior Scale, 2nd Edition (Vineland-II) | 3 years
  Standard assessment measuring communication, socializing, and daily living skills to assess their overall adaptive functioning for individuals up to 90 years of age. A higher score generally corresponds with higher adaptive function.
Caregiver Global Impression of Change (CaGI-C) | 3 years
  The CaGI-C is a caregiver reported outcome measure designed to assess any change in the subject's presentation over the preceding 7 days, as compared to the previous visit.

CONTACTS AND LOCATIONS:
Overall Officials: Elise Beausoleil, Study Director — Neurogene Inc.
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States